CLINICAL TRIAL: NCT05972109
Title: Multi-Level Trial of a Workplace Sales Ban of Sugary Beverages and Brief Motivational Counseling Intervention on Adiposity
Brief Title: Metabolic Health Improvement Program: Effects of a Workplace Sugary Beverages Sales Ban and Motivational Counseling
Acronym: MHIP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Sutter Health (Other); California Pacific Medical Center Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 22-38247; R01DK132870 (NIH)
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Obesity, Abdominal; Insulin Sensitivity
MeSH Terms: conditions — Obesity, Abdominal; Insulin Resistance | interventions — Crisis Intervention

STUDY DESIGN:
Intervention Model Description: The study is a double-randomized, controlled trial of 700 Sutter Health employees working at 16 hospital campuses. The hospital campuses will be randomized to sales ban or control. After screening employees at the 16 campuses for heavy SSB consumption (> 30 oz/week), the investigators will further randomize study participants to receive the brief counseling intervention or not. This will result in a balanced design of n=175 participants in each cell of a 2x2 factorial design: 1) sales ban alone; 2) behavioral counseling alone, 3) combined condition of sales ban and behavioral counseling, and 4) no intervention or control condition. This is an efficient design for testing the effects of the sales ban and brief counseling interventions plus their cross-level interaction within a context of full randomization.
Masking Description: The study is a double-randomized, controlled trial of 700 Sutter Health employees working at 16 hospital campuses. The hospital campuses will be randomized to sales ban or control. After screening employees at the 16 campuses for heavy SSB consumption (> 30 oz/week), the investigators will further randomize study participants to receive the brief counseling intervention or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control: No workplace SSB sales ban, no brief intervention (No Intervention): Participants receive no workplace SSB sales ban (environmental intervention) and no brief counseling intervention.
- Workplace SSB sales ban only (Experimental): Participants receive a workplace SSB sales ban (environmental intervention). This entails the removal of SSBs from all workplace sales outlets, replacing them with non-sugary beverage options.
  Interventions: Other: Workplace SSB sales ban
- Brief intervention only (Experimental): Participants receive a 20-30 minute intervention by video call, with 2 booster telephone calls. One week and one month after the initial session, participants will have 10-minute check-in/booster phone calls.
  Interventions: Behavioral: Brief Intervention
- Multilevel Intervention (workplace SSB sales ban + brief intervention) (Experimental): Sales ban: Participants receive a workplace SSB sales ban (environmental intervention). This entails the removal of SSBs from all workplace sales outlets, replacing them with non-sugary beverage options.
  Brief Intervention: Participants receive a 20-30 minute intervention by video call, with 2 booster telephone calls. One week and one month after the initial session, participants will have 10-minute check-in/booster phone calls.
  Interventions: Other: Workplace SSB sales ban; Behavioral: Brief Intervention

INTERVENTIONS:
Other: Workplace SSB sales ban — Environmental Intervention. The hospital food services will replace sugary drinks with non-sugar added alternative beverages throughout the campus.
  Arms: Multilevel Intervention (workplace SSB sales ban + brief intervention); Workplace SSB sales ban only
Behavioral: Brief Intervention — Participants receive single-session brief intervention, which is an intervention that uses motivational interviewing, and helps participants understand amount and effect of their baseline SSB intake, identify realistic goals for reduction and overcoming obstacles.
  Arms: Brief intervention only; Multilevel Intervention (workplace SSB sales ban + brief intervention)

SUMMARY:
The purpose of the study is to test the impact of a multilevel workplace intervention (hospital-wide sales ban on sugar-sweetened beverages (SSBs) and individual-level brief counseling) on employee health.

DETAILED DESCRIPTION:
This double-randomized controlled trial of a multilevel workplace intervention that combines an employer-sponsored sales ban on sugar-sweetened beverages (SSBs) with brief counseling to support reduced consumption will test how well each intervention works alone, whether they work better in combination than separately, and whether or not changes in SSB cravings mediate these effects. Sutter Health worksites will be randomly assigned to either a control condition or to implement a sales ban on SSBs. Within all sites, employees will be randomized to receive/not receive a brief counseling intervention focused on reducing SSB consumption. Participants will complete self-report questionnaires, give blood samples, and provide measurements of waist circumference, height, and weight. These data will be analyzed to determine the effects of the interventions, both separately and in combination.

ELIGIBILITY:
Inclusion Criteria:

* Full-time employee who works on campus at one of the Sutter Health participating sites
* Speaks and reads English
* Consumes three or more sugar-sweetened beverages (SSB) a week
* Agrees to participate in two fasting blood draws

Exclusion Criteria:

* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Abdominal Adiposity (Waist Circumference) | Baseline and 12 Months
  Waist circumference in centimeters (using method from Multi-Ethnic Study of Atherosclerosis). The study will measure the change between baseline and 12 month Abdominal Adiposity measurements.
Change in Insulin Sensitivity (HOMA) | Baseline and 12 Months
  Insulin sensitivity will be calculated using the homeostatic model assessment (HOMA). The equation for HOMA is fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5. The study will measure the change between baseline and 12 month HOMA.

SECONDARY OUTCOMES:
Change in Body Mass Index (BMI) | Baseline and 12 Months
  Body Mass Index [BMI] measured using height in centimeters and weight in kilograms to be calculated into BMI. The study will measure the change between baseline and 12 month BMI.
Change in Quantity of SSB Consumption | Baseline and 12 Months
  Fluid ounces of SSB consumed per day using Automated Self-Administered Dietary Assessment Tool (ASA-24) and Beverage Intake Questionnaire (BEV-Q). The study will measure the change between baseline and 12 month SSB consumption quantity.
Change in Lipid Profile Measurements | Baseline and 12 Months
  HDL, LDL, total cholesterol, triglycerides, and triglycerides:HDL ratio (calculated). The study will measure the change between baseline and 12 month individual lipid profile measurements (E.g., HDL, LDL, total cholesterol, triglycerides, and triglycerides:HDL ratio).
Change in ApoB Levels | Baseline and 12 Months
  Blood level of ApoB. The study will measure the change between baseline and 12 month ApoB blood levels.
Change in Fasting insulin Levels | Baseline and 12 Months
  Fasting blood level of insulin. The study will measure the change between baseline and 12 month Fasting insulin blood levels.
Change in Fasting Glucose Levels | Baseline and 12 Months
  Fasting blood level of glucose. The study will measure the change between baseline and 12 month Fasting Glucose blood levels.

OTHER OUTCOMES:
Change in Uric Acid Levels | Baseline and 12 Months
  Blood level of Uric Acid. The study will measure the change between baseline and 12 month Uric Acid blood levels.
Change in HbA1C Levels | Baseline and 12 Months
  Blood Level of HbA1C. The study will measure the change between baseline and 12 month HbA1C blood levels.

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Schmidt, Ph.D, Principal Investigator — University of California, San Francisco; Elissa Epel, Ph.D, Principal Investigator — University of California, San Francisco; Jamey Schmidt, Principal Investigator — Sutter Health/California Pacific Medical Center Research Institute
Locations (1):
- Sutter Health/California Pacific Medical Center Research Institute, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT05972109/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT05972109/ICF_001.pdf